CLINICAL TRIAL: NCT01774903
Title: Evaluation Study of Efficacy and Safety of TTS-Fentanyl in Severe Chronic Low Back Pain
Brief Title: An Efficacy and Safety Study of Transdermal Therapeutic System (TTS)-Fentanyl in Severe Chronic Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014533; FENPAI4051
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Results first posted 2013-03-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-02

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; TTS-fentanyl; Durogesic
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TTS-fentanyl (Experimental)
  Interventions: Drug: TTS-fentanyl

INTERVENTIONS:
Drug: TTS-fentanyl — TTS-fentanyl patches releasing drug at the rate of 12.5 microgram (µg) per hour for 3 days. The patches will be replaced every 3 days until 30 days.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Transdermal Therapeutic System (TTS)-fentanyl patch (transdermal patch containing a drug that is put on the skin so the drug will enter the body through the skin) in severe (very serious, life threatening) chronic (lasting a long time) low back pain in Thai participants.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention), single arm, prospective (study following participants forward in time) study conducted to assess the efficacy and safety of TTS-fentanyl in Thai participants with chronic low back pain. All participants start treatment with 12.5 micrograms (µg) per hour patch. The patches will be replaced every 3 days. On Day 3, and every 3 days thereafter, the TTS-fentanyl dose increases will be considered based on rescue medication consumption and pain assessment. No increase in TTS-fentanyl dose will be performed within the 72-hour dosing interval. The duration of the treatment will be 30 days. Primary efficacy assessment will be pain control rated by participants. Assessment time points will be at Day 0 (baseline), on Day 15 and Day 30 (trial end). At the end of study, global preference on efficacy, side effects and overall satisfaction will also be rated by investigator and participants. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria: -Chronic low back pain with moderate to severe pain at least 3 months -Participants needed to be treated with strong opioid and haven't been treated with strong opioid in the past -Participants who still had moderate to severe pain (Visual Analog Scale [VAS] >= 4), which was not adequately controlled by weak opioids such as tramadol or codeine at optimal doses (at least 120 milligram [mg] per day for tramadol or 200 mg per day for codeine) for at least 7 consecutive days

-Participants who failed from other treatments such as operation or lack of efficacy of current treatment -Participant who has signed the informed consent form Exclusion Criteria: -Skin disease that prevent the use of the transdermal system or which could affect the absorption of fentanyl or local tolerability -History or suspicion of alcohol or drug abuse within the past 5 years -History of cardiac, nervous system or respiratory disease which in the investigator's judgment precludes participation in the study because of the potential for respiratory depression -Concomitant use of Non Steroidal Anti-Inflammatory Drugs (NSAIDs), Cyclooxygenase - 2 (COX-2), muscle relaxant, topical analgesic during the previous week (unless on stable drug dose for at least 1 month before study entry) -Pregnancy or breast-feeding female; female participants of childbearing potential without adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (1):
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Transdermal Therapeutic System (TTS)-Fentanyl: TTS-fentanyl patches releasing at the rate of 12.5 microgram (mcg) per hour for 3 days. The patches were replaced every 3 days until 30 days.
Period: Overall Study
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Started | 45
Completed | 34
Not Completed | 11
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 1
Not completed — Ineligible to continue the trial | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Number analyzed (Participants) | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 55.80 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 13
Pain Intensity Score by Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: centimeter (cm)] — Assessed by 10 cm VAS from 0 to 10, where 0 cm=no pain and 10 cm=worse pain.
  centimeter (cm) | 6.57 (1.44)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity at Day 15
Description: Pain control was assessed by using a 10 centimeter (cm) visual analog scale (VAS) ranging from 0 to 10, where 0 cm=no pain and 10 cm=worse pain.
Time Frame: Day 15
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study medication and had at least one post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Number analyzed (Participants) | 37
cm | 4.85 (2.13)

2. Primary Outcome: Pain Intensity at Day 30
Description: Pain control was assessed by using a 10 cm VAS ranging from 0 to 10, where 0 cm=no pain and 10 cm=worse pain.
Time Frame: Day 30
Population: ITT population included all participants who received at least 1 dose of study medication and had at least one post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- TTS-fentanyl: TTS-fentanyl patches releasing at the rate of 12.5 microgram (mcg) per hour for 3 days. The patches were replaced every 3 days until 30 days.
Arm/Group | TTS-fentanyl
Number analyzed (Participants) | 37
cm | 4.89 (2.46)

3. Secondary Outcome: Number of Participants With Investigator Global Assessment
Description: Investigator completed a global assessment of the participants treatment with respect to pain control using a 9-point scale (-4 to 4; where, -4=100 percent worse, 0=unchanged and 4=100 percent improvement), safety using 5-point scale (1 to 5; where, 1=no, 2=mild, 3=moderate, 4=severe and 5=most severe side effects) and 5-point overall satisfaction scale (1-5; where, 1=no, 2=mild, 3=moderate, 4=good, 5=excellent).
Time Frame: Day 30
Population: Per protocol (PP) population included all participants who completed the 30-day study.
Measure: Number; unit: participants
Arm/Group | TTS-fentanyl
Number analyzed (Participants) | 34
participants
  Efficacy, 100 percent worse | 0
  Efficacy, 75 percent worse | 1
  Efficacy, 50 percent worse | 2
  Efficacy, 25 percent worse | 1
  Efficacy, unchanged | 6
  Efficacy, 25 percent improvement | 6
  Efficacy, 50 percent improvement | 11
  Efficacy, 75 percent improvement | 6
  Efficacy, 100 percent improvement | 1
  Safety, no | 17
  Safety, mild | 15
  Safety, moderate | 1
  Safety, severe | 1
  Safety, most severe | 0
  Overall satisfaction, no | 6
  Overall satisfaction, mild | 8
  Overall satisfaction, moderate | 11
  Overall satisfaction, good | 7
  Overall satisfaction, excellent | 2

4. Secondary Outcome: Number of Participants With Participant Global Assessment
Description: Participants completed a global assessment with respect to pain control using a 9-point scale (-4 to 4; where, -4=100 percent worse, 0=unchanged and 4=100 percent improvement), safety using 5-point scale (1 to 5; where, 1=no, 2=Mild, 3=Moderate, 4=Severe and 5=most severe side effects) and 5-point overall satisfaction scale (1-5; where, 1=no, 2=mild, 3=moderate, 4=good, 5=excellent).
Time Frame: Day 30
Population: PP population included all participants who completed the 30-day study.
Measure: Number; unit: participants
Arm/Group | TTS-fentanyl
Number analyzed (Participants) | 34
participants
  Efficacy, 100 percent worse | 1
  Efficacy, 75 percent worse | 0
  Efficacy, 50 percent worse | 2
  Efficacy, 25 percent worse | 1
  Efficacy, unchanged | 4
  Efficacy, 25 percent improvement | 13
  Efficacy, 50 percent improvement | 11
  Efficacy, 75 percent improvement | 1
  Efficacy, 100 percent improvement | 1
  Safety, no | 12
  Safety, mild | 15
  Safety, moderate | 6
  Safety, severe | 0
  Safety, most severe | 1
  Overall satisfaction, no | 3
  Overall satisfaction, mild | 10
  Overall satisfaction, moderate | 15
  Overall satisfaction, good | 5
  Overall satisfaction, excellent | 1

ADVERSE EVENTS:
Time Frame: From signing of informed consent until 30 days after the participant has completed the study
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl
Serious Adverse Events (participants affected / at risk) | 1/45
Other Adverse Events (participants affected / at risk) | 37/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transdermal Therapeutic System (TTS)-Fentanyl (N=45)
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Vertigo (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transdermal Therapeutic System (TTS)-Fentanyl (N=45)
Vomiting (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 17
Bitter taste (Nervous system disorders) | 1
Drowsiness (Nervous system disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Loss of appetizer (Metabolism and nutrition disorders) | 2
Palpitation (Cardiac disorders) | 2
Irritate (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Company has the right to publish the data which generated here under by Principal Investigator (PI), without PIs approval. The PI has the right to publish the results, but prior to submission, PI will provide at least 60 days to company for review. No paper that incorporates Company Confidential Information will be submitted for publication without Company prior written consent. If requested, the PI will withhold such publication for up to an additional 60 days to allow for filing of a patent.